CLINICAL TRIAL: NCT03850067
Title: A Phase 1b, Multicenter, Open-label, Dose Finding Study to Assess the Safety, Tolerability, and Preliminary Efficacy of CC-90011 Given in Combination With Cisplatin and Etoposide in First Line, Extensive Stage Subjects With Small Cell Lung Cancer
Brief Title: A Safety, Tolerability and Preliminary Efficacy Evaluation of CC-90011 Given in Combination With Cisplatin and Etoposide in Subjects With First Line, Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90011-SCLC-001; U1111-1228-2067 (Registry Identifier: WHO); 2018-002799-42 (EudraCT Number)
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Safety; CC-90011; Extensive stage small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pulrodemstat besilate; Cisplatin; Carboplatin; Etoposide; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CC-90011 in combination with Cisplatin and Etoposide (Experimental): During the Chemotherapy Treatment Period, the dose escalation is designed to explore three dose levels of CC-90011, for example 20, 40, and 60 mg as determined by Bayesian design, administered orally Days 1 and 8, in combination with cisplatin intravenous (IV) 75 mg/m2, Day 1, and etoposide iv 100 mg/m2 on Days 1, 2, and 3, for 4 cycles of 21 days each. Subjects completing the chemotherapy and being responders as per RECIST 1.1 will enter the Maintenance Treatment Period. Subjects completing 6 cycles of maintenance treatment subject will be treated only with CC-90011 at RP2D (60 mg) and continuing on CC-90011 are only required to have clinic visits/assessments performed on Day 1 (± 3 days) of each subsequent cycle (Cycles 6 and higher) unless more frequent visits are clinically indicated.
  Interventions: Drug: CC-90011; Drug: Cisplatin
- CC-90011 in combination with Carboplatin and Etoposide (Experimental): During the Chemotherapy Treatment Period, the dose escalation is designed to explore three dose levels of CC-90011, for example 20, 40, and 60 mg as determined by Bayesian design, administered orally Days 1 and 8, in combination with cisplatin intravenous (IV) 75 mg/m2, Day 1, and etoposide iv 100 mg/m2 on Days 1, 2, and 3, for 4 cycles of 21 days each. Subjects completing the chemotherapy and being responders as per RECIST 1.1 will enter the Maintenance Treatment Period. Subjects completing 6 cycles of maintenance treatment subject will be treated only with CC-90011 at RP2D (60 mg) and continuing on CC-90011 are only required to have clinic visits/assessments performed on Day 1 (± 3 days) of each subsequent cycle (Cycles 6 and higher) unless more frequent visits are clinically indicated
  Interventions: Drug: Carboplatin; Drug: Etoposide
- Nivolumab combination (Experimental): When the RP2D of CC-90011 in combination with cisplatin or carboplatin and etoposide is determined, the combination of CC-90011 at RP2D with cisplatin or carboplatin and etoposide plus nivolumab IV 240 mg Day 1 of each chemotherapy cycle, will be explored. For CC-90011 in combination with chemotherapy and nivolumab, the starting dose will be the RP2D of CC-90011 in combination with chemotherapy.
  A maintenance therapy will be given to subjects responding to the combination of CC-90011 with chemotherapy or to chemotherapy with nivolumab, as per RECIST 1.1. These subjects will receive 60 mg or 40 mg (in case of combination with nivolumab) of CC-90011 orally once weekly on Days 1, 8, 15, and 22, during cycles of 28-day each and, in the case of the combination with nivolumab, nivolumab IV 480 mg on Day 1 during cycles of 28-day each.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: CC-90011 — CC-90011
  Arms: CC-90011 in combination with Cisplatin and Etoposide
Drug: Cisplatin — Cisplatin
  Arms: CC-90011 in combination with Cisplatin and Etoposide
Drug: Carboplatin — Carboplatin
  Arms: CC-90011 in combination with Carboplatin and Etoposide
Drug: Etoposide — Etoposide
  Arms: CC-90011 in combination with Carboplatin and Etoposide
Drug: Nivolumab — Nivolumab
  Arms: Nivolumab combination

SUMMARY:
CC-90011-SCLC-001 is a multicenter, Phase 1b, open-label, dose finding study to assess the safety, tolerability, and preliminary efficacy of CC-90011 given concurrently and sequentially to standard of care platinum-based, cisplatin and etoposide, carboplatin and etoposide and/or etoposide and Nivolumab to subjects with first line ES SCLC.

The dose finding part of the study will explore escalating oral doses of CC-90011 in combination with cisplatin, etoposide and/or carboplatin with or without Nivolumab (chemotherapy), to determine the maximum tolerated dose of CC- 90011 in combination with chemotherapy with or without Nivolumab to subjects with first line ES SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subject is 18 years of age or older at the time of signing the informed consent form (ICF).
2. Subject with histological or cytological confirmation of extensive stage SCLC according to 2015 WHO classification (Travis, 2015).
3. Subject must be able to provide fresh or archival tumor tissues
4. Subject is found suitable for at least 4 cycles of platinum-based standard chemotherapy.
5. Subject has at least 1 site of measurable disease per RECIST 1.1.
6. Subject must have the following laboratory values:

   • Absolute neutrophil count (ANC) ≥ 1.5 x 109/L

   • Hemoglobin (Hgb) ≥ 10 g/dL (≥ 100 g/L or > 6.2 mmol/L)
   * Platelet count (Plt) ≥ 150 x 109/L
   * Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamate pyruvate transaminase (ALT/SGPT) ≤ 3.0 x upper limit of normal (ULN) or ≤ 5.0 x ULN if liver metastases are present
   * Serum total bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 60 mL/min (see Appendix G to see creatinine clearance formula). For the purposes of this protocol, the glomerular filtration rate (GFR) is considered to be equivalent to the creatinine clearance.
   * Prothrombin time (or international normalized ratio [INR]) and activated partial thromboplastin time (APTT) ≤ 1.5 ULN
7. Females of childbearing potential (FCBP) must:

   • Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use one highly effective contraceptive method plus one barrier method.
   * Have two negative pregnancy tests as verified by the Investigator prior to starting CC-90011:

     - a negative serum pregnancy test (sensitivity of at least 25 mIU/mL) at Screening

     - a negative serum or urine pregnancy test within 24 hours prior to Cycle 1 Day 1 of study treatment.

     - a negative Serum or urine within 24 hours prior to first dose of nivolumab and then every 4 weeks (± 1 week) regardless of dosing schedule.
   * Avoid conceiving for 6 months after last dose of cisplatin or carboplatin or etoposide, or 5 months after last dose of nivolumab for FCBP, or 45 days after the last dose of CC-90011, whichever is the latest.
   * Agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
8. Males must practice true abstinence from heterosexual intercourse (which must be reviewed on a monthly basis) or agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or an FCBP and will avoid conceiving from signing the ICF, while participating in the study, during dose interruptions, and for 6 months after last dose of cisplatin, or carboplatin, or etoposide or at least 105 days following CC-90011 discontinuation, whichever is the latest, even if he has undergone a successful vasectomy.
9. Males must agree to refrain from donating sperm while on treatment and females must agree to refrain from donating ova while on treatment and for 6 months after the last dose of cisplatin or etoposide or 105 days after last dose of CC-90011.
10. Subject is able to swallow pills.

Exclusion Criteria:

1. Subject has received anticancer therapy (either approved or investigational, including radiation with curative intent) for SCLC prior to study entry.
2. Subject has undergone major surgery ≤ 4 weeks prior to Cycle 1 Day 1 or has not recovered from surgery.
3. Subject has persistent diarrhea due to a malabsorptive syndrome (such as celiac sprue or inflammatory bowel disease) ≥ NCI CTCAE Grade 2, despite medical management), or any other significant gastrointestinal (GI) disorder that could affect the absorption of CC- 90011.
4. Subject with symptomatic or uncontrolled ulcers (gastric or duodenal), particularly those with a history of and/or risk of perforation and GI tract hemorrhages.
5. Subject with any hemorrhage/bleeding event > CTCAE Grade 2 or hemoptysis > 1 teaspoon within 4 weeks prior to the first dose.
6. Subject with symptomatic and untreated or unstable central nervous system (CNS) metastases.
7. Subject has impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   - Left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition (MUGA) scan or echocardiogram (ECHO).

   - Complete left bundle branch or bifascicular block.

   - Congenital long QT syndrome.

   - Persistent or clinically meaningful ventricular arrhythmias or atrial fibrillation.

   - QTcF ≥ 480 msec on Screening ECG (mean of triplicate recordings).
8. Subject has other clinically significant heart disease such as congestive heart failure requiring treatment or uncontrolled hypertension (blood pressure ≥ 160/95 mm Hg).
9. Subject is a pregnant or nursing female.
10. Subject has known human immunodeficiency virus (HIV) infection.
11. Subject has known chronic active hepatitis B or C virus (HBV, HCV) infection.
12. Subject with ongoing treatment with chronic, therapeutic dosing of anticoagulants (eg, warfarin, low molecular weight heparin, Factor Xa inhibitors, thrombin antagonist).
13. Subject has a history of concurrent second cancers requiring active, ongoing systemic treatment.
14. Subject has Grade 2 peripheral sensory neuropathy.
15. Subject with poor bone marrow reserve as assessed by Investigator.
16. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
17. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
18. Previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to C1D1.

    • Acute symptoms must have resolved and based on investigator assessment in consultation with the medical monitor, there are no sequelae that would place the participant at a higher risk of receiving study treatment
19. Previous SARS-CoV-2 vaccine within 7 days of C1D1. For vaccines requiring more than one dose, the full series (e.g. both doses of a two-dose series) should be completed prior to C1D1 when feasible and when a delay in C1D1 would not put the study subject at risk
20. Subject has any condition that confounds the ability to interpret data from the study.

    For the subjects treated with nivolumab:
21. Subject has received prior therapies targeting PD-1 or PD-L1
22. Subject has a history of persistent skin rash ≥ NCI CTCAE Grade 2.
23. Subject with an autoimmune disease, or any other condition, requiring systemic treatment with either corticosteroids within 14 days (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 30 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

    * Subjects with type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

22. Subject has received treatment with botanical preparations (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks prior to randomization. Refer to Section 8.2 for prohibited therapies.

23. Subject has history of allergy or hypersensitivity to study drug components.

24. Subject has received a live/attenuated vaccine within 30 days of first treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to approximately 2 years
  A DLT is defined as any of the toxicities described in the protocol occurring within the DLT assessment unless the event can clearly be determined to be unrelated to CC-90011
Maximum Tolerated Dose (MTD) | Up to approximately 2 years
  MTD is the highest dose that causes DLTs in not more than 33% of the subjects treated with CC-90010 in the first cycle with at least 6 evaluable subjects treated at this dose
Adverse Events (AEs) | Up to approximately 3 years
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
  Is defined as the percent of subjects whose best response is complete response (CR) or partial response (PR).
Progression-free Survival (PFS) | Up to approximately 2 years
  Is defined as the time from the first dose of study drug to the first occurrence of disease progression or death from any cause.
Overall Survival (OS) | Up to approximately 2 years
  Is measured as the time from the first dose of CC-90011 to death due to any cause.
Pharmacokinetics- Cmax | Up to approximately 2 years
  Maximum observed plasma concentration
Pharmacokinetics- AUC | Up to approximately 2 years
  Area under the plasma concentration time-curve
Pharmacokinetics- Tmax | Up to approximately 2 years
  Time to maximum plasma concentration
Pharmacokinetics- t1/2 | Up to approximately 2 years
  Terminal half-life
Pharmacokinetics- CL/F | Up to approximately 2 years
  Apparent clearance
Pharmacokinetics- VzF | Up to approximately 2 years
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb; Oscar Juan Vidal, MD, PhD, Principal Investigator — Hospital Universitario La Fe; Stefania Salvagni, MD, Principal Investigator — Azienda Ospedaliero Universitarua, Policlinico S. Orsola Malpighi; Rossana Berardi, MD, Principal Investigator — Ospedali Riuniti di Ancona; Armando Santoro, MD, Principal Investigator — IRCCS Instituto Clinic Humanitas; Benjamin Besse, MD, PhD, Principal Investigator — Gustave Roussy, Ditep
Locations (13):
- France (3):
  - Local Institution - 102, Marseille
  - Local Institution - 103, Saint-Herblain
  - Local Institution - 100, Villejuif
- Italy (3):
  - Local Institution - 203, Ancona
  - Local Institution - 200, Bologna
  - Local Institution - 201, Rozzano (MI)
- Spain (7):
  - Local Institution - 406, Majadahonda, Madrid
  - Local Institution - 403, Barcelona
  - Local Institution - 402, Barcelona
  - Local Institution - 400, Madrid
  - Local Institution - 404, Málaga
  - Local Institution - 405, Valencia
  - Local Institution - 401, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Kanouni T, Severin C, Cho RW, Yuen NY, Xu J, Shi L, Lai C, Del Rosario JR, Stansfield RK, Lawton LN, Hosfield D, O'Connell S, Kreilein MM, Tavares-Greco P, Nie Z, Kaldor SW, Veal JM, Stafford JA, Chen YK. Discovery of CC-90011: A Potent and Selective Reversible Inhibitor of Lysine Specific Demethylase 1 (LSD1). J Med Chem. 2020 Dec 10;63(23):14522-14529. doi: 10.1021/acs.jmedchem.0c00978. Epub 2020 Oct 9. PMID 33034194
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT03850067.html